CLINICAL TRIAL: NCT07403838
Title: The Impact of Preoperative Chronic Pain on Postoperative Depressive States in Elderly Patients Undergoing Joint Replacement Surgery: A Secondary Analysis Based on Prospective Data
Status: Completed | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: The Affiliated Hospital Of Guizhou Medical University (Other)
Responsible Party: Principal Investigator, Weidong Mi, Director of the Department of Anesthesiology, The First Medical Center of Chinese PLA General Hospital, Chinese PLA General Hospital
Other Study IDs: PLAGH-PSD-001
Record Dates: First submitted 2026-02-01; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Postoperative Depression
Keywords: Postoperative Depression Chronic Pain Elderly Patients Joint Replacement; Postoperative Depressive Symptoms; Postoperative Acute Pain; Preoperative Chronic Pain; Elderly
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background:

Postoperative depression is a significant complication that hinders recovery in elderly patients undergoing joint replacement surgery. Although preoperative chronic pain is common in this population and pain and depression frequently coexist, the predictive role and underlying mechanisms of preoperative chronic pain on postoperative depression remain unclear. This study aims to systematically explore the association between the two, providing a basis for optimizing perioperative management and improving patient outcomes.

Methods:

This study is a secondary analysis of multicenter prospective data, including elderly patients who underwent elective knee or hip replacement surgery between April 2020 and April 2022 from a perioperative database of elderly patients in China. The impact of preoperative chronic pain on the occurrence of depressive states within 7 days after surgery was systematically evaluated using univariate and multivariate logistic regression analysis, propensity score matching, and subgroup analysis.

DETAILED DESCRIPTION:
Introduction Against the backdrop of the deepening global trend of population aging, the number of elderly individuals undergoing joint replacement surgery has increased significantly. Although this surgery effectively alleviates pain and restores joint function, perioperative mood disorders have become a key factor affecting patient recovery and long-term quality of life [1]. Among common orthopedic surgeries in the elderly, hip and knee replacements hold a prominent position. Since joint function directly impacts patients' basic living abilities such as walking and mobility, the risk of postoperative anxiety and depression is particularly pronounced. Studies indicate that the incidence of depression after joint replacement surgery can reach 33%, while the incidence of anxiety ranges between 25% and 33% [2,3]. Preoperative chronic pain is a prevalent clinical symptom in this patient population; however, whether an association exists between it and postoperative depression remains unclear due to a lack of systematic clinical evidence.

Notably, elderly patients undergoing joint replacement often have a long history of chronic pain, with studies showing a preoperative pain prevalence as high as 43.2% [4]. Known common risk factors for depression in the elderly include gender, age, sleep status, pain, and activities of daily living [5-7]. In the perioperative context, studies have confirmed that postoperative pain exacerbates mood disorders and increases the prevalence of depression [4]. However, compared to postoperative pain, preoperative chronic pain may exert multifaceted effects on postoperative outcomes, including mood and functional recovery [4,8]. Pre-existing chronic pain, as a potential and important predictor, has not been sufficiently explored for its unique impact on postoperative depression.

Based on this background, this study included 575 elderly patients undergoing joint replacement surgery to investigate the effect of preoperative chronic pain on postoperative depression in this population.

II. Research Objectives and Significance

Objectives:

To investigate the impact of preoperative chronic pain on postoperative depressive states in elderly patients undergoing joint replacement surgery, providing evidence to optimize perioperative management, reduce depression risk, and improve patient outcomes.

Significance:

Postoperative depression increases complications and adversely affects prognosis in elderly patients. By analyzing the impact of preoperative chronic pain on postoperative depressive states in elderly joint replacement patients, this study provides evidence to support interventions aimed at reducing postoperative depression. Addressing preoperative chronic pain may help prevent the occurrence of postoperative depressive states in elderly patients undergoing joint replacement surgery.

**III. Research Content** The correlation between preoperative chronic pain and postoperative depressive states in elderly patients undergoing joint replacement surgery. This study is a retrospective cohort study based on prospectively collected data. It extracts relevant data from the Perioperative Database of Elderly Patients in China for patients aged 65 and older who underwent joint replacement surgery between April 2020 and April 2022. Patients were divided into a no-chronic-pain group and a chronic-pain group based on the presence of preoperative chronic pain. Perioperative data were statistically analyzed to observe the occurrence of depressive states within one week postoperatively, as well as postoperative hospital stay length, postoperative acute pain, anxiety symptoms within one week, and the incidence of delirium.

IV. Study Design

1. This study is a retrospective cohort study based on prospectively collected data.

   Sample Size:A post-hoc power analysis was performed using G*Power 3.1 software. Parameters were set as: significance level (α) two-tailed = 0.05, sample size (N) = 575. The results indicated that for correlation analysis (point-biserial correlation), this sample size is sufficient to achieve over 99% power (1-β) to detect an effect size (correlation coefficient r) as low as 0.1. This power far exceeds the commonly accepted standard of 80% in academia [9]. Therefore, the final inclusion of 575 patients in our study is adequate.

   Study Groups:Patients were divided into two groups based on the exposure factor (presence of preoperative chronic pain): Group 1: No chronic pain group; Group 2: Chronic pain group.

   Target Population:The data for this study were sourced from the Perioperative Database of Elderly Patients in China. This is a prospective observational cohort study conducted across multiple centers, which prospectively collected perioperative data from patients aged 65 and older undergoing elective non-cardiac, non-neurosurgical surgery at 19 tertiary hospitals between April 1, 2020, and April 30, 2022. This study is a secondary analysis of this database and will retrospectively extract the following existing data from eligible patients who underwent elective joint replacement surgery during the same period: (1) Baseline characteristics: age, gender, body mass index (BMI), American Society of Anesthesiologists physical status (ASA) classification, smoking, alcohol use, preoperative chronic pain history, comorbidities (hypertension, diabetes, coronary heart disease, cerebrovascular disease, hepatic insufficiency, renal insufficiency); (2) Preoperative laboratory tests (most recent before surgery): hemoglobin (Hb), white blood cell count, serum albumin; (4) Intraoperative variables: operation duration, bleeding and transfusion, intraoperative medications (dexmedetomidine, opioids, non-steroidal anti-inflammatory drugs, inhaled anesthetics), anesthesia method, and use of drainage tubes and analgesic pumps.

   Exposure Factor:The presence of preoperative chronic pain.
2. Primary and Secondary Outcomes Primary Outcome: Occurrence of depressive states within 7 days postoperatively. Secondary Outcomes: Incidence of anxiety states within 7 days postoperatively; incidence of delirium within 7 days postoperatively; postoperative hospital stay length; incidence of postoperative acute pain.

   Postoperative Depressive State: Assessed at bedside within 7 days postoperatively by uniformly trained researchers using the Chinese version of the Patient Health Questionnaire-9 (PHQ-9). A PHQ-9 score >5 was defined as the occurrence of a depressive state [10].

   Postoperative Anxiety State: Assessed at bedside within 7 days postoperatively by uniformly trained researchers using the Chinese version of the Generalized Anxiety Disorder-7 (GAD-7) scale. A GAD-7 score >5 was defined as the occurrence of an anxiety state [11].

   Delirium:Assessed at bedside within 7 days postoperatively by uniformly trained researchers using the Chinese version of the 3D-CAM scale. Assessments were conducted twice daily, in the morning and afternoon. The Chinese version of the 3D-CAM scale is a widely adopted and validated assessment tool [12].

   Postoperative Pain: Assessed using the Numerical Rating Scale (NRS). An NRS score ≥4 on the first postoperative day was defined as the occurrence of moderate-to-severe acute pain [13].
3. Statistical Analysis Models were established based on the collected perioperative indicators. Univariate and multivariate logistic regression analyses, propensity score matching, and subgroup analyses were employed to explore the impact of preoperative chronic pain on postoperative depressive states.

V. Participant Inclusion/Exclusion Criteria and Withdrawal/Discontinuation Criteria

Clinical data were retrospectively included for patients aged 65 years and older who underwent joint replacement surgery between April 2020 and April 2022 from the Perioperative Database of Elderly Patients in China.

Inclusion Criteria:

1. Age ≥ 65 years.
2. No cognitive impairment, defined as a preoperative Mini-Mental State Examination (MMSE) score below the education-adjusted cutoff: ≤17 points for illiterate individuals, ≤20 points for those with incomplete primary education, and ≤23 points for those with incomplete junior high school education.
3. Underwent elective joint replacement surgery.
4. Completed postoperative assessments, including questionnaires for depression, anxiety, and delirium.

Exclusion Criteria:

1. Non-general anesthesia.
2. Patients admitted to the intensive care unit postoperatively.
3. Medical centers with fewer than 50 cases.

Data were collected strictly according to the inclusion and exclusion criteria.

**VI. Management Plan for Common/Serious Adverse Reactions**

This study is a retrospective cohort study and does not involve adverse reactions resulting from experimentation.

VII. Statistical Methods

Normally distributed continuous variables are expressed as mean ± standard deviation (SD) and compared using t-tests. If continuous data are not normally distributed, they are presented as median and interquartile range (IQR) and compared using the Mann-Whitney test. Categorical variables are expressed as frequencies or percentages and compared using the χ2 test or Fisher's exact test. Statistical significance was set at the 0.05 level, and all tests were two-tailed. Logistic regression models were performed using R version 4.0.1.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 65 years.
2. No cognitive impairment or history of mental illness.
3. Underwent elective joint replacement surgery.
4. Completed postoperative assessments, including questionnaires for depression, anxiety, and delirium.

Exclusion Criteria:

1. Non-general anesthesia.
2. Patients admitted to the intensive care unit postoperatively.
3. Medical centers with fewer than 50 cases. -

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: This study is a secondary analysis based on a multicenter prospective database. We included 881 elderly patients who underwent elective joint replacement surgery at multiple medical centers between April 2020 and April 2022. The data were sourced from the Perioperative Database of Elderly Patients in China, which is a multicenter prospective study. The primary aim of this parent study was to identify perioperative risk factors in elderly patients undergoing non-cardiac surgery and to establish a targeted risk prevention and management system, utilizing data collected over a two-year period from 19 hospitals across the nation.
Sampling Method: Non-Probability Sample
Enrollment: 575 (Actual)
Dates: Start 2022-04-30 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Incidence and Severity Classification of Postoperative Depressive States (within 7 days) | within 7 days after surgery
  Postoperative depressive states were assessed using the Chinese version of the Patient Health Questionnaire-9 (PHQ-9). This scale was administered at bedside within 7 days after surgery by trained researchers. It is a self-reported tool comprising 9 items and is widely used for the efficient screening of clinical depressive symptoms. The assessment results were interpreted as follows: a total score ≥ 5 indicated the presence of a postoperative depressive state, with scores of 5-9 classified as mild, 10-14 as moderate, and 15-27 as moderately severe to severe.

CONTACTS AND LOCATIONS:
Overall Officials: Li TONG TONG, PHD, Principal Investigator — Department of Anesthesiology, The First Medical Center of Chinese PLA General Hospital; Weidong MI Mi, PHD, Study Director — Department of Anesthesiology, The First Medical Center of Chinese PLA General Hospital
Locations (1):
- Department of Anesthesiology, First Medical Center of the People's Liberation Army General Hospital, Beijing, Haidian, China

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) generated in this study are not planned to be shared publicly. The data contain sensitive personal health information and are subject to confidentiality protections under the ethical approval and data management regulations governing this research. Data access is restricted to the immediate research team for the purposes outlined in the approved study protocol

REFERENCES:
- [Result] Li L, Wu P, Wang Z, Meng X, Zha C, Li Z, Qi T, Zhang Y, Han B, Li S, Jiang C, Zhao Z, Cai J. NoncoRNA: a database of experimentally supported non-coding RNAs and drug targets in cancer. J Hematol Oncol. 2020 Feb 28;13(1):15. doi: 10.1186/s13045-020-00849-7. PMID 32111231
- [Result] Ninova M, Ronshaugen M, Griffiths-Jones S. Conserved temporal patterns of microRNA expression in Drosophila support a developmental hourglass model. Genome Biol Evol. 2014 Aug 27;6(9):2459-67. doi: 10.1093/gbe/evu183. PMID 25169982
- [Result] Thomson KH, Rantala MH, Viita-Aho TK, Vainio OM, Kaartinen LA. Condition-based use of antimicrobials in cats in Finland: results from two surveys. J Feline Med Surg. 2009 Jun;11(6):462-6. doi: 10.1016/j.jfms.2008.10.005. Epub 2008 Dec 25. PMID 19111491
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/39837610/